CLINICAL TRIAL: NCT02721823
Title: Randomized Controlled Trial on the Effect of Stress Reduction and Lifestyle Modification on Disease Activity in Ulcerative Colitis
Brief Title: Randomized Controlled Trial of Stress Reduction and Lifestyle Modification for Ulcerative Colitis
Acronym: MBMCol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Jost Langhorst, Medical vice director, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-6554-BO
Record Dates: First submitted 2016-02-10; First posted 2016-03-29 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- lifestyle-modification (Experimental): Once a week for 10 weeks with a circumference of 60 hours with mindfulness-based stress reduction and further process of the Mind / body medicine.
  Interventions: Behavioral: lifestyle-modification
- control group (Active Comparator): A unique education unit within the scope of 3 hours on the influence of lifestyle factors on the disease and self-help materials for the independent training.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: lifestyle-modification — The group intervention is carried out once a week for 10 weeks for a total of 60 hours with elements of mindfulness-based stress reduction (MBSR) and further process of the mind / body medicine. In this project, this program will be adapted to the specific needs of colitis patients.
  Arms: lifestyle-modification
Behavioral: Control group — Participants in this group receive a one-time education unit within the scope of 3 hours on the influence of lifestyle factors on the disease, also self-help materials for independent training offered. Following the follow-up measure also this group is given the opportunity to participate in the multimodal stress reduction- and lifestyle modification program.
  Arms: control group

SUMMARY:
Patients with ulcerative colitis often suffer significant limitations to their quality of life, which are also conditioned by particular stress and psychosocial accompanying symptoms of the disease. A multimodal program for stress-reduction and lifestyle-modification has been shown to be effective in promoting the quality of life. The study will examine the promotion of the quality of life of patients with ulcerative colitis and the positive Influence on stress, psychological symptoms and physiological parameters. 92 patients with ulcerative colitis will be randomized in an Intervention group and a control group for 10 weeks. The primary outcome is the disease-specific quality of life, the secondary outcomes are stress, psychological symptoms, inflammatory parameters, disease activity parameters, bowel parameter and the microbiome.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years
* diagnosis of ulcerative colitis
* Currently in remission, remission not longer than 12 months
* limited quality of life or increased subjective stress level

Exclusion Criteria:

* Infectious or chronic active ulcerative colitis
* Taking glucocorticoids or immunosuppressants within the last 3 months, except stable medication using azathioprine
* colectomy
* serious psychological disorder (for example: major depression, addiction, schizophrenia)
* serious comorbid somatic disease (for example: diabetes mellitus, oncological disease)
* pregnancy
* participation in stress reduction program or clinical studies to psychological interventions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Disease-specific quality of life | 12 weeks
  Inflammatory Bowel Disease Questionnaire (IBD-Q)

SECONDARY OUTCOMES:
Disease-specific quality of life | 48 weeks
  Inflammatory Bowel Disease Questionnaire (IBD-Q)
Disease-specific quality of life | 60 weeks
  Inflammatory Bowel Disease Questionnaire (IBD-Q)
Disease-specific quality of life | 108 weeks
  Inflammatory Bowel Disease Questionnaire (IBD-Q)
Disease activity | 12 weeks
  Mayo Disease Activity Index (Mayo Score)
Disease activity | 12 weeks
  Clinical Activity Index (CAI)
Disease activity | 48 weeks
  Mayo Disease Activity Index (Mayo Score)
Disease activity | 48 weeks
  Clinical Activity Index (CAI)
Disease activity | 60 weeks
  Mayo Disease Activity Index (Mayo Score)
Disease activity | 60 weeks
  Clinical Activity Index (CAI)
Disease activity | 108 weeks
  Mayo Disease Activity Index (Mayo Score)
Disease activity | 108 weeks
  Clinical Activity Index(CAI)
Endoscopic index | 12 weeks
  Endoscopic-Index (sigmoidoscopy)
Endoscopic index | 48 weeks
  Endoscopic-Index (sigmoidoscopy)
Endoscopic index | 60 weeks
  Endoscopic-Index (sigmoidoscopy))
Endoscopic index | 108 weeks
  Endoscopic-Index (sigmoidoscopy)
Histology | 12 weeks
  Riley Score
Histology | 48 weeks
  Riley Score
Histology | 60 weeks
  Riley Score
Histology | 108 weeks
  Riley Score
Generic quality of life | 12 weeks
  Short Form (SF) -36 (items) health survey
Generic quality of life | 48 weeks
  SF-36 health survey
Generic quality of life | 60 weeks
  SF-36 health survey
Generic quality of life | 108 weeks
  SF-36 health survey
Anxiety and depression | 12 weeks
  Hospital Anxiety and Depression Scale (HADS)
Anxiety and depression | 48 weeks
  Hospital Anxiety and Depression Scale (HADS)
Anxiety and depression | 60 weeks
  Hospital Anxiety and Depression Scale (HADS)
Anxiety and depression | 108 weeks
  Hospital Anxiety and Depression Scale (HADS)
Perceived stress | 12 weeks
  Perceived Stress Scale (PSS)
Perceived stress | 48 weeks
  Perceived Stress Scale (PSS)
Perceived stress | 60 weeks
  Perceived Stress Scale (PSS)
Perceived stress | 108 weeks
  Perceived Stress Scale (PSS)
Irritable Bowel Syndrome Symptoms | 12 weeks
  IBS Severity Scoring System (IBS-SSS)
Irritable Bowel Syndrome Symptoms | 48 weeks
  IBS Severity Scoring System (IBS-SSS)
Irritable Bowel Syndrome Symptoms | 60 weeks
  IBS Severity Scoring System (IBS-SSS)
Irritable Bowel Syndrome Symptoms | 108 weeks
  IBS Severity Scoring System (IBS-SSS)
Hemogram | 12 weeks
  leukocyte, hemoglobin, hematocrit, platelet
Hemogram | 48 weeks
  leukocyte, hemoglobin, hematocrit, platelet
Hemogram | 60 weeks
  leukocyte, hemoglobin, hematocrit, platelet
Hemogram | 108 weeks
  leukocyte, hemoglobin, hematocrit, platelet
Blood sedimentation rate | 12 weeks
Blood sedimentation rate | 48 weeks
Blood sedimentation rate | 60 weeks
Blood sedimentation rate | 108 weeks
C-reactive protein | 12 weeks
C-reactive protein | 48 weeks
C-reactive protein | 60 weeks
C-reactive protein | 108 weeks
faecal calprotectin | 12 weeks
faecal calprotectin | 48 weeks
faecal calprotectin | 60 weeks
faecal calprotectin | 108 weeks
faecal lactoferrin | 12 weeks
faecal lactoferrin | 48 weeks
faecal lactoferrin | 60 weeks
faecal lactoferrin | 108 weeks
faecal polymorphonuclear (PMN)-elastase | 12 weeks
  faecal polymorphonuclear elastase
faecal PMN-elastase | 48 weeks
  faecal polymorphonuclear elastase
faecal PMN-elastase | 60 weeks
  faecal polymorphonuclear elastase
faecal PMN-elastase | 108 weeks
  faecal polymorphonuclear elastase
faecal human beta-defensin-2 (hBD-2) | 12 weeks
faecal hBD-2 | 48 weeks
  human beta-defensin-2
faecal hBD-2 | 60 weeks
  human beta-defensin-2
faecal hBD-2 | 108 weeks
  human beta-defensin-2
Intestinal microbiota | 12 weeks
  High-throughput 16S ribosomal ribonucleic acid (rRNA) gene sequencing
Intestinal microbiota | 48 weeks
  High-throughput 16S rRNA gene sequencing
Intestinal microbiota | 60 weeks
  High-throughput 16S rRNA gene sequencing
Intestinal microbiota | 108 weeks
  High-throughput 16S rRNA gene sequencing
Intestinal permeability | 12 weeks
  LactoseMonitol
Intestinal permeability | 48 weeks
  LactoseMonitol
Intestinal permeability | 60 weeks
  LactoseMonitol
Intestinal permeability | 108 weeks
  LactoseMonitol
Adverse events | 12 weeks
Adverse events | 48 weeks
Adverse events | 60 weeks
Adverse events | 108 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jost Langhorst, Prof. Dr. med., Principal Investigator — Kliniken Essen-Mitte
Locations (1):
- Kliniken Essen-Mitte, Knappschafts Krankenhaus, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391
- [Derived] Schlee C, Uecker C, Bauer N, Koch AK, Langhorst J. Multimodal stress reduction and lifestyle modification program for patients with ulcerative colitis: a qualitative study. BMC Complement Med Ther. 2022 Mar 8;22(1):60. doi: 10.1186/s12906-021-03478-w. PMID 35260152